CLINICAL TRIAL: NCT05417529
Title: Preoperative Music Listening Versus Intravenous Midazolam (PMLOS) on Anxiety, Sedation and Stress in Odontostomatological Surgery: a Randomized Controlled Study
Brief Title: Preoperative Music Listening in Odontostomatological Surgery (PMLOS)
Acronym: PMLOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MTI.ODONTO
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Stage I or II Micro-invasive Oral Cancer
Keywords: music therapy; stress; sedation; surgery; anesthesia
MeSH Terms: interventions — Reference Standards

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatement Group (Experimental): Participants received music therapy intervention
  Interventions: Other: music therapy intervention
- Control Group (Active Comparator): Patients in control group receive premedication
  Interventions: Drug: Standard Preparation

INTERVENTIONS:
Other: music therapy intervention — Participants did not receive premedication with midazolam 0,02 mg/kg intravenous and received music therapy intervention by a certified music therapist FAMI . Music Treatment consisted of 3 steps:
  (1)30 minutes before surgery, music therapist (MTp) engaged the patient in an individual brief conversation (10 min.) to identify preferred musical genre/songs and prepared a customized playlists to listen to during induction; (2)After being monitored in the operating room, patients were prepared to listening to music ; (3)Music listening during anesthesia induction. Anesthesia was the same in both groups. Induction was carried out by fentanyl 3mcg/kg, propofol 2 mg/kg and rocuronium at the dose of 1mg/kg to facilitate intubation
  Arms: Treatement Group
Drug: Standard Preparation — Partecipants receive premedication with midazolam 0,02 mg/kg intravenous. Anesthesia was the same in both groups. Induction was carried out by fentanyl 3mcg/kg, propofol 2 mg/kg and rocuronium at the dose of 1mg/kg to facilitate intubation
  Arms: Control Group

SUMMARY:
People undergoing general anesthesia for oral cancer diagnosis and treatment often experience heightened anxiety, fear and stress with negative bodily responses, such as tachycardia, hypertension, increased myocardial consumption of O2, arrhythmias, increased peripheral resistance, hypercoagulability, immunodeficiency and catabolic response . Emotional distress and pain may be managed by pre-procedurally application of anxiolytic, analgesic, and anesthetic drugs, but with potential risks or side effects such as respiratory depression, nausea and vomiting, confusion, memory loss, hypoxemia, and drug-drug interactions. This may result in adverse outcomes, such as delayed healing, increased healthcare utilization, and cost.

A recent Cochrane review showed that benzodiazepines reduce pre-procedural anxiety compared with placebo with a low quality of evidence.

Music therapy (MT), defined as the clinical and evidence-based use of music interventions by a trained professional for the purpose of achieving individualized goals within a therapeutic relationship between patient, music and music therapist 6 , may be used as a safe and cost-effective complementary intervention in adjunct to standard surgical care.

During surgery, music is a powerful positive stimulus that evokes and modulates emotions as well as mood, face mask adverse stimuli, and improves emotional health through coping.

Music therapy and music medicine interventions are effective to prevent and treat emotional distress and pain before, during and after medical procedures .

Evidence from Cochrane systematic reviews shows that music interventions affect positively anxiety in patients with cancer, coronary heart diseases and in patients on mechanical ventilation .

Some studies reported also that music interventions reduced sedative requirements in patients undergoing surgery under regional anesthesia combined with sedation, both with midazolam and propofol and also in critically ill patients in intensive care units.

The primary aim of this study was to evaluate the effects of preoperative music therapy intervention compared to premedication with midazolam on anxiety, sedation and stress during general anesthesia for odontostomatological elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* no severe neurological or psychiatric conditions,
* no hearing impairment,
* no drugs abuse,
* American Society of Anesthesiologists (ASA) score I to III

Exclusion Criteria:

* < 18 years
* severe neurological or psychiatric conditions,
* hearing impairment,
* drugs abuse,
* American Society of Anesthesiologists (ASA) score IV to V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | 30 minutes before
  Anxiety Visual Analogues Scale (A-VAS) was used to evaluate the level of anxiety from 0 (no anxiety) to 10 (maximum anxiety) before surgical procedure T0
Anxiety | 60 minutes after
  Anxiety Visual Analogues Scale (A-VAS) was used to evaluate the level of anxiety from 0 (no anxiety) to 10 (maximum anxiety) before surgical procedure T0
Bispectral Index (BIS) | during anesthesia induction
  Bispectral index (BIS) is one of several technologies used to monitor depth of anesthesia. BIS monitors are used to supplement Guedel's classification system for determining depth of anesthesia. Titrating anesthetic agents to a specific bispectral index during general anesthesia in adults (and children over 1 year old) allows the anesthetist to adjust the amount of anesthetic agent to the needs of the patient, possibly resulting in a more rapid emergence from anesthesia.
  BIS monitoring is widely used in clinical anesthesia as an index for monitoring the electrical activity of the cerebral cortex and the sedative ingredients of anesthesia. BIS scores range from 0 to 100 (0, coma; 40-60, general anesthesia; 60-90, sedated; 100, awake) and reflect the level of sedation regardless of a patient's clinical characteristics or the type of sedative drug used.
Patient global impression of satisfaction (PGIS) | through study completion, 1 hour after surgery
  Patient global impression of satisfaction (PGIS) with a 4 items score ( 1=very dissatisfied, 2=dissatisfied, 3=satisfied, 4=very satisfied).

SECONDARY OUTCOMES:
Blood Pressure (SBP-DPB) | during the procedure
Heart Rate | during the procedure
O2SAT | during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Filomena Puntillo, PhD, Principal Investigator — University of Bari
Locations (1):
- AOUC Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koelsch S, Fuermetz J, Sack U, Bauer K, Hohenadel M, Wiegel M, Kaisers UX, Heinke W. Effects of Music Listening on Cortisol Levels and Propofol Consumption during Spinal Anesthesia. Front Psychol. 2011 Apr 5;2:58. doi: 10.3389/fpsyg.2011.00058. eCollection 2011. PMID 21716581
- [Result] Marcantonio ER, Juarez G, Goldman L, Mangione CM, Ludwig LE, Lind L, Katz N, Cook EF, Orav EJ, Lee TH. The relationship of postoperative delirium with psychoactive medications. JAMA. 1994 Nov 16;272(19):1518-22. PMID 7966844
- [Result] Ebrahimi R, Shroyer AL, Dennis P, Currier J, Lendvai Wischik D. Music Can Reduce the Need for Pharmacologic Conscious Sedation During Invasive Coronary Angiography. J Invasive Cardiol. 2020 Nov;32(11):440-444. doi: 10.25270/jic/20.00132. Epub 2020 Oct 22. PMID 33087584
- [Result] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Result] Chlan LL, Heiderscheit A, Skaar DJ, Neidecker MV. Economic Evaluation of a Patient-Directed Music Intervention for ICU Patients Receiving Mechanical Ventilatory Support. Crit Care Med. 2018 Sep;46(9):1430-1435. doi: 10.1097/CCM.0000000000003199. PMID 29727366
- [Result] Palmer JB, Lane D, Mayo D, Schluchter M, Leeming R. Effects of Music Therapy on Anesthesia Requirements and Anxiety in Women Undergoing Ambulatory Breast Surgery for Cancer Diagnosis and Treatment: A Randomized Controlled Trial. J Clin Oncol. 2015 Oct 1;33(28):3162-8. doi: 10.1200/JCO.2014.59.6049. Epub 2015 Aug 17. PMID 26282640
- [Result] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797
- [Result] Ortega A, Gauna F, Munoz D, Oberreuter G, Breinbauer HA, Carrasco L. Music Therapy for Pain and Anxiety Management in Nasal Bone Fracture Reduction: Randomized Controlled Clinical Trial. Otolaryngol Head Neck Surg. 2019 Oct;161(4):613-619. doi: 10.1177/0194599819856604. Epub 2019 Jun 11. PMID 31184266
- [Result] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Result] Fallek R, Corey K, Qamar A, Vernisie SN, Hoberman A, Selwyn PA, Fausto JA, Marcus P, Kvetan V, Lounsbury DW. Soothing the heart with music: A feasibility study of a bedside music therapy intervention for critically ill patients in an urban hospital setting. Palliat Support Care. 2020 Feb;18(1):47-54. doi: 10.1017/S1478951519000294. PMID 31104642
- [Result] Giordano F, Losurdo A, Quaranta VN, Campobasso N, Daleno A, Carpagnano E, Gesualdo L, Moschetta A, Brienza N. Effect of single session receptive music therapy on anxiety and vital parameters in hospitalized Covid-19 patients: a randomized controlled trial. Sci Rep. 2022 Feb 24;12(1):3154. doi: 10.1038/s41598-022-07085-8. PMID 35210504
- [Result] Kertai MD, Whitlock EL, Avidan MS. Brain monitoring with electroencephalography and the electroencephalogram-derived bispectral index during cardiac surgery. Anesth Analg. 2012 Mar;114(3):533-46. doi: 10.1213/ANE.0b013e31823ee030. Epub 2012 Jan 17. PMID 22253267